CLINICAL TRIAL: NCT00639847
Title: A Randomized Controlled Study to Evaluate the Role of an In Home Asthma Disease Management Program Provided by Respiratory Therapists in Improving Outcomes and Reducing the Cost of the Care
Brief Title: This Study Compared an in Home Asthma Management Program Provided by Nurses or Respiratory Therapist
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Jay Peters, MD, University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 989-0030-090
Record Dates: First submitted 2008-03-13; First posted 2008-03-20 (Estimated); Last update posted 2008-03-24 (Estimated); Status verified 2008-03

CONDITIONS: Asthma
Keywords: Asthma management; cost; disease management; respiratory care; nursing; health care utilization; health related quality of life
MeSH Terms: conditions — Asthma; Patient Acceptance of Health Care | interventions — Adenosine Monophosphate

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- group 1 (No Intervention): this is the standard of care control group. The control group will be instructed to return to their regular physicians for routine follow up at a time to be specified by the physician.
- Group 2 (Active Comparator): Group 2 will receive routine home visits from nurses provided by a home health care agency.
  Interventions: Behavioral: In-home asthma management program (AMP) provided by nurses
- Group 3 (Active Comparator): In-home asthma management program (AMP) provided by respiratory therapists. The AMP included asthma education (medications use, monitoring, triggers, steps to manage asthma attacks), demonstration and training (peak flow meter use, MDI and nebulizer use, asthma diary), home environment assessment and suggestions for environmental changes (mattress covers, control of dust, pets, fumes, cleaning materials, cock roach control, etc.)
  Interventions: Behavioral: In-home asthma management program (AMP) provided by respiratory therapists

INTERVENTIONS:
Behavioral: In-home asthma management program (AMP) provided by nurses — The AMP included asthma education (medications use, monitoring, triggers, steps to manage asthma attacks), demonstration and training (peak flow meter use, MDI and nebulizer use, asthma diary), home environment assessment and suggestions for environmental changes (mattress covers, control of dust, pets, fumes, cleaning materials, cock roach control, etc.)
  Arms: Group 2
Behavioral: In-home asthma management program (AMP) provided by respiratory therapists — The AMP included asthma education (medications use, monitoring, triggers, steps to manage asthma attacks), demonstration and training (peak flow meter use, MDI and nebulizer use, asthma diary), home environment assessment and suggestions for environmental changes (mattress covers, control of dust, pets, fumes, cleaning materials, cock roach control, etc.)
  Arms: Group 3

SUMMARY:
This study compared an in-home asthma management program provided by nurses or respiratory therapists to see if those receiving program had fewer hospitalizations, clinic and emergency room visits and higher levels of satisfaction and health related quality of life.

DETAILED DESCRIPTION:
Background: Disease management may improve outcomes and reduce cost. We compared an in-home asthma management program (AMP) delivered by respiratory therapists (RTs) or nurses (RNs) to standard care (SC) in 159 adults with moderate to severe asthma to determine the effect on health care utilization (HCU), patient satisfaction (PS) and health related quality of life (HRQOL).

Methods: This single center, prospective trial randomized subjects, age 18-64, to three groups: SC, AMP-RT or AMP-RN. Outcomes at six-months were HCU, cost, pulmonary function, symptoms, environmental assessment, asthma self-management, HRQOL (SF-36; St. Georges Respiratory Questionnaire [SGRQ]) and PS. Frequencies were compared using chi 2; all other variables were compared using ANOVA with a post-hoc test.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 18-64 years) treated in the ED or hospitalized for an acute exacerbation of asthma at the university teaching hospital were invited to participate.

Exclusion Criteria:

* Included other pulmonary disorders or diagnosis of co-morbid disease which was disabling in nature.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 159 (Actual)
Dates: Start 1998-10; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Health care utilization (hospitalizations, hospital days, emergency room visits, clinic visits) and cost. | 6 months

SECONDARY OUTCOMES:
Health related quality of life (SF-36 and St. George's Respiratory Questionnaire), oxygenation, pulmonary function, symptoms, patient satisfaction and asthma self-management score | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David C Shelledy, PhD, Principal Investigator — University of Texas; Terry S. Le Grand, PhD, Principal Investigator — University of Texas; Donna D. Gardner, MSHP, Principal Investigator — University of Texas; Jay I Peters, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States